CLINICAL TRIAL: NCT03768219
Title: Phase 1 Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of APVO210 in Healthy Subjects, Patients With Psoriasis, and Patients With Ulcerative Colitis
Brief Title: Study to Evaluate APVO210 in Healthy Subjects, Patients With Psoriasis, and Patients With Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8001
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Psoriasis; Ulcerative Colitis
MeSH Terms: conditions — Psoriasis; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: SAD: Randomized, double-blind, placebo-controlled, sequential cohort-group study with a sentinel subject design
  MAD: Randomized, double-blind, placebo-controlled, sequential cohort-group study
  Psoriasis Expansion Cohort: Randomized, double-blind, placebo-controlled study
  Ulcerative Colitis Expansion Cohort: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Stage 1 (SAD) Cohort 1 (Experimental): 6 subjects will receive 2 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 2 (Experimental): 6 subjects will receive 5 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 3 (Experimental): 6 subjects will receive 10 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 4 (Experimental): 6 subjects will receive 20 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 5 (Experimental): 6 subjects will receive 40 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 6 (Experimental): 6 subjects will receive 80 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 7 (Experimental): 6 subjects will receive 160 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 1 (SAD) Cohort 8 (Experimental): 6 subjects will receive 320 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 2 (MAD) Cohort 9 (Experimental): 8 subjects will receive 40 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 2 (MAD) Cohort 10 (Experimental): 8 subjects will receive 80 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 2 (MAD) Cohort 11 (Experimental): 8 subjects will receive 160 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Stage 2 (MAD) Cohort 12 (Experimental): 8 subjects will receive 360 mcg/kg of APVO210 2 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Expansion Cohort (Psoriasis) (Experimental): 12 subjects will receive the starting dose for the Psoriasis Patients Expansion Cohort portion of the study will be the recommended dose from Stage 2 of the study of APVO210. It will be a dose that has been demonstrated to be safe and well tolerated by the Safety Monitoring Committee.
  8 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo
- Expansion Cohort (Ulcerative Colitis) (Experimental): 12 Subjects will receive the starting dose for the Ulcerative Colitis Patients Expansion Cohort portion of the study will be the recommended dose from Stage 2 of the study of APVO210. It will be a dose that has been demonstrated to be safe and well tolerated by the Safety Monitoring Committee.
  8 subjects will receive placebo
  Interventions: Biological: APVO210; Biological: Placebo

INTERVENTIONS:
Biological: APVO210 — APVO210
Biological: Placebo — Placebo is saline based IV infusion, and is identical in appearance to active study drug.

SUMMARY:
Phase 1 study in 2 stages with 2 expansion cohorts. The first stage is a single ascending dose (SAD) study of APVO210 in healthy volunteers. The second stage is a multiple ascending dose (MAD) study of APVO210 in healthy volunteers. Two expansion cohorts evaluate multiple doses of APVO210 in psoriasis patients and ulcerative colitis patients.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

* Age 18 to 65 years old.
* Body mass index (BMI) > 18.5 kg/m2 and < 30.0 kg/m2; minimum body weight of 50 kg.
* Good health and no clinically significant findings on:
* Physical examination
* 12-lead ECG
* Clinical laboratory tests (serum chemistry, haematology, coagulation, urine drug screen, and urinalysis (UA))
* Seated systolic blood pressure (BP) 90 to 140 mm Hg.
* Seated diastolic BP 60 to 90 mm Hg.

Psoriasis Patients (Expansion Cohort):

Main Inclusion Criteria:

* Clinical diagnosis of chronic plaque psoriasis with a disease duration of at least 6 months; patients with concurrent psoriatic arthritis may be enrolled.
* Psoriasis Area and Severity Index (PASI) score ≥ 12 at baseline.
* Psoriasis plaque BSA (Body surface area) ≥ 10%
* PGA (Physician Global Assessment) ≥ 3.
* Age 18 to 65 years old.
* Body mass index > 18.5 and < 35.0 kg/m2; minimum body weight of 50 kg.

Ulcerative Colitis Patients (Expansion Cohort):

Main Inclusion Criteria:

* Moderately to severely active ulcerative colitis as defined by:
* Baseline Mayo Score of 6 to 12; and
* Endoscopic sub-score ≥2 as read by central reader
* Is intolerant, refractory, or only partially responsive to corticosteroids (not including budesonide), immunomodulators (azathioprine [AZA] or 6-mercaptopurine [6-MP], and methotrexate), or biologics.
* Age 18 to 65 years old.
* Body mass index > 18.5 and < 35.0 kg/m2; minimum body weight of 50 kg.

Exclusion Criteria:

Main Exclusion Criteria

* Clinically significant manifestation of metabolic; hepatic; renal; haematological; pulmonary; cardiovascular; gastrointestinal; musculoskeletal; dermatological; urogenital; eye, ear, nose, and throat; psychiatric; or neurological disorders.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.2 times the upper limit of normal (ULN) as defined by the laboratory.
* Positive hepatitis panel (hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV]) or positive human immunodeficiency virus (HIV) antibody.
* Positive Quantiferon tuberculosis (TB) test at Screening Visit.
* Receipt of live vaccine less than 1 month prior to Check in or plan to receive live vaccine during the study or up to 3 months following End of Treatment visit.
* Infection in the 4 weeks prior to Check-in that required hospitalization or parenteral antibiotics.

Psoriasis Patients (Expansion Cohort):

Main Exclusion Criteria:

* History of malignancy, diagnosed or known to be active or actively treated within the past 5 years, other than resected lesions of low malignant potential, such as basal cell skin cancers or low risk squamous cell carcinomas of the skin.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN) as defined by the laboratory.
* Creatinine > 1.5 times ULN as defined by the laboratory.
* Positive hepatitis panel (hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV]) or positive human immunodeficiency virus (HIV) antibody.
* Positive Quantiferon tuberculosis (TB) test at Screening Visit.
* Receipt of live vaccine less than 1 month prior to Check in or plan to receive live vaccine during the study or up to 3 months following End of Treatment visit.
* Infection in the 4 weeks prior to Check-in that required hospitalization or parenteral antibiotics.
* Use of a prescription medication that could have an effect on psoriasis (eg, lithium, systemic steroids, immunosuppressants) during the 14 days before Check-in; use of prescription medications for psoriasis is not permitted until after the Follow-up Visit.
* Non plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular).
* Use of biologic agents (eg, adalimumab, etanercept, infliximab, ustekinumab, ixekizumab, secukinumab, guselkumab, tildrakizumab, brodalumab) or psoralen and ultraviolet A (PUVA) within 12 weeks prior to Check-in, ultraviolet B (UVB) phototherapy, use of tanning beds, or use of systemic medications such as methotrexate, cyclosporine A, acitretin, tofacitinib or apremilast within 4 weeks prior to Check-in, or topical anti-psoriasis medications (except emollients) within 2 weeks prior to Check-in.

Ulcerative Colitis Patients (Expansion Cohort):

Main Exclusion Criteria:

* Ulcerative colitis requiring immediate surgical, endoscopic, or radiological intervention including massive haemorrhage, perforation and sepsis, suppurative complications, or toxic colon.
* Stool positive for Clostridium difficile toxin, enteric pathogens, or ova and parasites.
* Positive hepatitis panel (hepatitis B surface antigen [HBsAg] and anti hepatitis C virus [HCV]) or positive human immunodeficiency virus (HIV) antibody.
* Positive Quantiferon tuberculosis (TB) test at Screening Visit.
* Receipt of live vaccine less than 1 month prior to Check in or plan to receive live vaccine during the study or up to 3 months following End of Treatment visit.
* Infection in the 4 weeks prior to Check-in that required hospitalization or parenteral antibiotics.
* Use of biologic agents (eg, adalimumab, etanercept, infliximab, ustekinumab, ixekizumab, secukinumab, guselkumab, tildrakizumab, brodalumab) or psoralen and ultraviolet A (PUVA) within 12 weeks prior to Check-in, ultraviolet B (UVB) phototherapy, use of tanning beds, or use of systemic medications such as methotrexate, cyclosporine A, acitretin, tofacitinib or apremilast within 4 weeks prior to Check-in, or topical anti-psoriasis medications (except emollients) within 2 weeks prior to Check-in.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to Day 29
Number of subjects with clinically relevant findings in vital signs | up to Day 29
Number of subjects with significant changes from baseline laboratory measurements | up to Day 29
Number of subjects with clinically significant abnormalities in electrocardiogram (ECG) results | up to Day 29
Number of subjects with clinical significant abnormalities found on physical examination | up to Day 29
Number of subjects with adverse events | up to Day 57
Number of subjects with clinically relevant findings in vital signs | up to Day 57
Number of subjects with significant changes from baseline laboratory measurements | up to Day 57
Number of subjects with clinically significant abnormalities in electrocardiogram (ECG) results | up to Day 57
Number of subjects with clinical significant abnormalities found on physical examination | up to Day 57
Number of psoriasis patients with adverse events | up to day 141
Number of psoriasis patients with clinically relevant findings in vital signs | up to day 141
Number of psoriasis patients with significant changes from baseline laboratory measurements | up to day 141
Number of psoriasis patients with clinically significant abnormalities in electrocardiogram (ECG) results | up to day 141
Number of psoriasis patients with clinical significant abnormalities found on physical examination | up to day 141
Number of ulcerative colitis patients with adverse events | up to day 141
Number of ulcerative colitis patients with clinically relevant findings in vital signs | up to day 141
Number of ulcerative colitis patients with significant changes from baseline laboratory measurements | up to day 141
Number of ulcerative colitis patients with clinically significant abnormalities in electrocardiogram (ECG) results | up to day 141
Number of ulcerative colitis patients with clinical significant abnormalities found on physical examination | up to day 141

SECONDARY OUTCOMES:
The number of subjects who develop anti-drug antibodies to APVO210 | Up to day 29
The number of subjects who develop anti-drug antibodies to APVO210 | Up to day 57
The number of psoriasis patients who develop anti-drug antibodies to APVO210 | Up to day 141
The number of ulcerative colitis patients who develop anti-drug antibodies to APVO210 | Up to day 141
Serum level of Peak Plasma Concentration (Cmax) | Up to day 29
Serum level of Peak Plasma Concentration (Cmax) | Up to day 57
Serum level of Peak Plasma Concentration (Cmax) in psoriasis patients | Up to day 141
Serum level of Peak Plasma Concentration (Cmax) in ulcerative colitis patients | Up to day 141
Area under the plasma concentration versus time curve (AUC) | Up to day 29
Area under the plasma concentration versus time curve (AUC) | Up to day 57
Area under the plasma concentration versus time curve (AUC) for psoriasis patients | Up to day 141
Area under the plasma concentration versus time curve (AUC) for ulcerative colitis patients | Up to day 141
Change in number of leukocytes by flow cytometry in psoriasis patients | Up to day 141
Change in number of leukocytes by flow cytometry in ulcerative colitis patients | Up to day 141
Change in cytokine levels by ex-vivo LPS stimulation assay in psoriasis patients. | Up to day 141
Change in cytokine levels by ex-vivo LPS stimulation assay in ulcerative colitis patients. | Up to day 141

CONTACTS AND LOCATIONS:
Overall Officials: David Schaaf, MD, Principal Investigator — Aptevo Therapeutics
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No